CLINICAL TRIAL: NCT06068153
Title: A Multicentre, Single-arm Phase II Trial of Sotorasib Plus Lenvatinib, As Second-line Treatment in Patients with KRASG12C-mutant, Metastatic NSCLC
Brief Title: AMG510 (sotorasib) Plus Lenvatinib As Second-line Treatment in Patients with KRASG12C Mutant, Metastatic NSCLC
Acronym: AMBER
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: In view of the recent developments in the field (the increasing number of trials with new KRAS inhibitors), the window of opportunity to answer the question raised in the AMBER trial was missed.
Sponsor: ETOP IBCSG Partners Foundation (Network)
Collaborators: Amgen (Industry); Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ETOP 24-22
Record Dates: First submitted 2023-09-28; First posted 2023-10-05 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Metastatic Non Small Cell Lung Cancer; KRAS G12C
Keywords: Metastatic NSCLC; KRAS G12C; Sotorasib; Lenvatinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — sotorasib; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm (Experimental): Sotorasib + Lenvatinib
  Interventions: Drug: Sotorasib; Drug: Lenvatinib

INTERVENTIONS:
Drug: Sotorasib — Sotorasib is administered at a dose of 960 mg (8x 120 mg) orally, once daily until progression or unacceptable toxicity.
Drug: Lenvatinib — Lenvatinib is administered at a dose of 20 mg orally (2x 10 mg), once daily until progression or unacceptable toxicity.

SUMMARY:
AMBER is a multicentre, single-arm phase II trial. The protocol treatment consists of of sotorasib plus lenvatinib, as a second-line treatment. The primary objective of the trial is to evaluate the clinical efficacy of sotorasib plus lenvatinib, in terms of objective response rate, for patients with KRASG12C-mutant, metastatic NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically documented metastatic NSCLC.
* Documented disease progression on prior treatment. Prior treatment must have included platinum-based doublet chemotherapy and immune-checkpoint inhibition.
* KRASG12C-mutation (identified through local molecular testing, using a validated test).
* Measurable disease per RECIST v1.1 criteria.
* Age ≥18 years.
* ECOG Performance Status of 0-1.
* Life expectancy of >3 months.
* Ability to swallow oral medications and willing to complete a treatment diary.
* Adequate haematological function.
* Adequate renal function.
* Adequate liver function.
* Men and women of childbearing potential must use highly effective contraception.
* Women of childbearing potential, including women who had their last menstruation in the last 2 years, must have a negative urinary or serum pregnancy test within 5 weeks before enrolment. Pregnancy test must be repeated within 3 days before the first dose of protocol treatment.
* Written IC for study participation must be signed and dated by the patient and the investigator prior to any study-related intervention.

Exclusion Criteria:

* Active brain metastases E.g., untreated brain lesions (new or progressing) and/or symptomatic brain lesions (symptoms as determined by the investigator).

Patients who have had brain metastases resected or have received whole brain radiation therapy ending at least 4 weeks (or stereotactic radiosurgery ending at least 2 weeks) prior to enrolment are eligible if they meet all of the following criteria:

* Residual neurological symptoms are only of grade ≤2
* On stable doses of dexamethasone or equivalent for at least 2 weeks, if applicable.
* History or presence of haematological malignancies. Exception: curatively treated haematological malignancies with no disease evidence in the last 2 years.
* History of (non-infectious) pneumonitis that required steroids or evidence of ILD/pneumonitis.
* Active hepatitis B and C and uncontrolled HIV.
* Uncontrolled blood pressure (systolic blood pressure >150 mmHg or diastolic blood pressure >90 mmHg) in spite of an optimised regimen of antihypertensive medication.
* Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, long QT syndrome (LQTS), unstable angina, myocardial infarction or stroke within 6 months before enrolment, or cardiac arrhythmia requiring medical treatment at screening
* Bleeding or thrombotic disorders or patients at risk for severe haemorrhage. The degree of tumour invasion/infiltration of major blood vessels (e.g. carotid artery) should be considered because of the potential risk of severe haemorrhage associated with tumour shrinkage/necrosis following lenvatinib therapy.
* Current or recent (within 10 days of enrolment) use of aspirin (>325 mg/day) or treatment with dipyramidole, ticlopidine, clopidogrel, or clostazol.
* Electrolyte abnormalities that have not been corrected.
* Proteinuria on urine dipstick testing >1+, unless a 24-hour urine collection for quantitative assessment indicates that the urine protein is <2 g/24 hours.
* History of abdominal or tracheoesophageal fistula or gastrointestinal perforation within 6 months prior to inclusion.
* Unresolved toxicities from previous lines of anti-cancer treatment regimens and/or (with the exception of alopecia) complications from major surgery prior to enrolment.
* Previous treatment with KRAS- and/or VEGF/R inhibitors.
* Hypersensitivity to sotorasib or lenvatinib.
* Women who are pregnant or breastfeeding or who are planning to become pregnant or breastfeed.
* Sexually active men and women of childbearing potential who are not willing to use a highly effective contraceptive method during the trial and for 7 days after the last dose of sotorasib and until 30 days after the last dose of lenvatinib.
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | From date of enrolment until 18 weeks post-enrolment.
  ORR is defined as the rate of patients, among all enrolled patients, achieving a best overall response [complete response (CR) or partial response (PR)] according to RECIST v1.1, investigator assessed, by 18 weeks post-enrolment.

SECONDARY OUTCOMES:
Progression-free survival per RECIST v1.1 | From the date of enrolment until last tumour assessment (approximately 22 months after the enrolment of the first patient)
  PFS is defined as the time from the date of enrolment until the date of documented progression (according to RECIST v1.1) or death from any cause, if progression is not documented. Censoring (for patients without progression or death) will occur at the date of last tumour assessment. Patients without a post-baseline tumour assessment will be censored at the date of enrolment plus 1 day.
Disease control rate per RECIST v1.1 | From date of enrolment until 18 weeks post-enrolment.
  DCR is defined as the rate of patients, among all enrolled patients, that achieve CR or PR or disease stabilisation (according to RECIST v1.1, investigator assessed) at 18 weeks.
Overall survival | From the date of enrolment until death from any cause (up to 22 months after the enrolment of the first patient)
  OS is defined as the time from the date of enrolment until the date of death from any cause. Censoring (for patients who are not reported as dead) will occur at the date last known to be alive. Data for patients who do not have post-baseline information will be censored at the date of enrolment plus 1 day.
Duration of response | From the date of enrolment until last tumour assessment or death from any cause (approximately 22 months after the enrolment of the first patient)
  DoR is defined as the interval from the date of first documentation of objective response (CR or PR, according to RECIST v1.1) to the date of first documented progression/relapse or death from any cause.
Adverse events according to CTCAE v5.0 | [Time Frame: From the date of enrolment until last patient last visit (approximately 22 months after enrolment of the first patient)]
  All safety parameters will be summarised in tables in order to evaluate the toxicity and safety profile of the protocol treatment based on:
  * Adverse events (AEs) according to CTCAE v5.0 (any-cause as well as treatment-related) including AEs leading to dose delays and/or interruptions, withdrawal of protocol treatment, and death
  * Severe, serious, and selected AEs
  * Deaths
  * Clinically significant laboratory parameters and abnormalities, and vital signs.

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Addeo, Study Chair — Département d'Oncologie Hôpitaux Universitaires de Genève; Sanjay Popat, Study Chair — Royal Marsden NHS Foundation Trust
Locations (15):
- Medical University of Innsbruck / UK für Innere Medizin V, Innsbruck, Austria
- University Hospital of Munich (LMU), Department of Medicine V (Pneumology/Thoracic Oncology), Munich, Germany
- Spain (8):
  - Alicante University Dr Balmis Hospital ISABIAL, Alicante
  - Ico Badalona - Hospital Germans Trias I Pujol, Badalona
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Nuestra Señora de Candelaria, Santa Cruz de Tenerife
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Universitario de Toledo, Toledo
  - Hospital Universitario Y Politécnico La Fe, Valencia
- Switzerland (5):
  - Istituto Oncologico della Svizzera Italiana, Bellinzona
  - Kantonsspital Graubünden, Chur
  - HFR Fribourg, Fribourg
  - HUG, Geneva
  - Kantonsspital Winterthur, Winterthur

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP